CLINICAL TRIAL: NCT04079452
Title: Doravirine Concentrations and Antiviral Activity in Cerebrospinal Fluid in HIV-1 Infected Individuals
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Collaborators: Institut d'Investigació Biomèdica de Bellvitge (Other); Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, Daniel Podzamczer, PhD: chief of the HIV and STD Unit (Infectious Disease Service), Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DORACeNeS; 2018-003915-24 (EudraCT Number)
Record Dates: First submitted 2019-09-03; First posted 2019-09-06 (Actual); Results first posted 2022-04-28 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: HIV-1-infection
Keywords: Doravirine
MeSH Terms: interventions — doravirine; emtricitabine tenofovir alafenamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Doravirine + Descovy® TAF/FTC (Experimental): Doravirine (MK-1439) 100 mg administered orally once daily in combination with Tenofovir alafenamide (TAF) and emtricitabine (FTC) coformulated as single tablet (Descovy® TAF/FTC 25/200 mg) and administered orally once daily during 4 weeks
  Interventions: Drug: Doravirine; Drug: Descovy

INTERVENTIONS:
Drug: Doravirine — Doravirine 100 mg tablet
  Other Names: MK-1439
Drug: Descovy — Tenofovir alafenamide 25 mg / emtricitabine 200 mg tablet
  Other Names: TAF/FTC

SUMMARY:
Doravirine is a new HIV-1 non-nucleoside reverse transcriptase inhibitor (NNRTI) that has demonstrated a good efficacy and safety profile in clinical trials. It functions by inhibiting viral replication of both wild-type virus and most common NNRTI variants. It is dosed orally once daily and always given in combination with other HIV-1 active agents as part of highly active antiretroviral therapy. Initial pharmacokinetic studies demonstrated not extensive binding to plasma proteins, which may be crucial determinant for penetration to different reservoirs such as the central nervous system (CNS). This study will address two important issues: The pharmacokinetic profile of Doravirine in cerebrospinal fluid (CSF) as well as the maintenance of HIV suppression in CSF. The assessment of concentrations as well as the antiviral activity of new antiretroviral drugs in compartments such as CNS is relevant to avoid HIV-related neurocognitive disorders as well as for future cure strategies. In addition, the role of unbound ARV drug concentrations has been scarcely evaluated.

DETAILED DESCRIPTION:
15 asymptomatic, virologically suppressed, HIV infected patients will be offered to switch their antiretroviral treatment to Doravirine+Emtricitabine/TAF. After 4 weeks of treatment all subjects will undergo lumbar puncture and bloods in order to assess CSF and plasma (total and unbound) Doravirine concentrations. HIV RNA also will be assessed. All subjects will complete a follow up visit 4 weeks after

ELIGIBILITY:
Inclusion Criteria:

1. Asymptomatic, HIV-1 infected individuals ≥ 18 years of age
2. Be on a stable ART continously or ≥3 consecutive months preceding the screening visit. Patients already receiving TAF/FTC+DoravirineC for at least three consecutive months will be eligible.
3. Plasma HIV-1 RNA at screening <40 copies/mL for at least 3 months at the Screening visit.
4. Signed and dated written informed consent prior to inclusion.
5. Subjects must agree to utilize a highly effective method of contraception during heterosexual intercourse from the screening visit throughout the duration of the study.

Exclusion Criteria:

1. Severe hepatic impairment (Child-Pugh Class C)
2. Ongoing malignancy
3. Active opportunistic infection
4. Primary resistance to any of the ARV included in the study or history of virologic failure with risk of resistance selection to any of the study drugs.
5. Any verified Grade 4 laboratory abnormality
6. ALT or AST ≥ 3xULN and/or bilirubin ≥ 1.5xULN
7. Adequate renal function: Estimated glomerular filtration rate ≥ 50 mL/min
8. Females who are pregnant (as confirmed by positive serum pregnancy test) or breastfeeding.
9. Current treatment with antiaggregant or anticoagulant therapy.
10. History of any neurologic disease/condition/treatment may alter the blood brain barrier permeability.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Podzamczer, PhD Chief, Principal Investigator — Hospital Universitari de Bellvitge
Locations (1):
- Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Doravirie+TAF/FTC Arm (Single Arm): Doravirine (100 mg)+ Tenofovir Alafenamide (TAF) and emtricitabine (FTC) co-formulated (TAF/FTC 25/200 mg)
Period: Overall Study
Arm/Group | Doravirie+TAF/FTC Arm (Single Arm)
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Doravirine + Descovy® TAF/FTC
Number analyzed (Participants) | 15
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 47 [27 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Spain | 15

OUTCOME MEASURES:

1. Primary Outcome: Total Doravirine Concentrations in Cerebrospinal Fluid
Description: Total Doravirine concentrations in cerebrospinal fluid in HIV-1 infected individual receiving ART with Doravirine+FTC/TAF
Time Frame: 4 Weeks
Population: Descriptive analysis was performed for all participants (15), defining median and IQR of Doravirine concentrations in CSF
Measure: Median (Inter-Quartile Range); unit: ng/ml
Groups:
- Doravirine+TAF/FTC Arm (Single Arm): Doravirine (100 mg)+ Tenofovir Alafenamide (TAF) and emtricitabine (FTC) co-formulated (TAF/FTC 25/200 mg)
Arm/Group | Doravirine+TAF/FTC Arm (Single Arm)
Number analyzed (Participants) | 15
ng/ml | 58.6 [23.2 to 127.3]

2. Primary Outcome: Total Doravirine Concentrations in Blood Plasma
Description: Total Doravirine concentrations in blood plasma
Time Frame: 4 Weeks
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Doravirie+TAF/FTC Arm (Single Arm)
Number analyzed (Participants) | 15
ng/ml | 417.6 [169.5 to 942.2]

3. Primary Outcome: Total Doravirine Concentration CSF/Plasma Ratio
Description: total Doravirine CSF/plasma ratio
Time Frame: 4 Weeks
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Doravirine+TAF/FTC Arm (Single Arm)
Number analyzed (Participants) | 15
ratio | 0.13 [0.09 to 0.19]

4. Primary Outcome: HIV-1 RNA in Cerebrospinal Fluid
Description: Number of patients with HIV-1 RNA cerebrospinal fluid <40 copies/ml
Time Frame: 4 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Doravirine+TAF/FTC Arm (Single Arm)
Number analyzed (Participants) | 15
Participants | 13

5. Primary Outcome: HIV-1 RNA in Blood Plasma
Description: Number of patients with HIV-1 RNA in blood plasma <40 copies/ml
Time Frame: 4 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Doravirine+TAF/FTC Arm (Single Arm)
Number analyzed (Participants) | 15
Participants | 14

6. Primary Outcome: Unbound Doravirine Concentrations in CSF
Description: Unbound Doravirine concentrations in cerebrospinal fluid in HIV-1 infected individual receiving ART with Doravirine+FTC/TAF
Time Frame: 4 Weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Doravirine+TAF/FTC Arm (Single Arm)
Number analyzed (Participants) | 15
ng/ml | 44.6 [14.9 to 105]

7. Primary Outcome: Doravirine Concentrations in Blood Plasma
Description: Unbound Doravirine concentrations in blood plasma
Time Frame: 4 Weeks
Measure: Median (Inter-Quartile Range); unit: CSF Unbound DORAVIRINE conc. ng/ml
Arm/Group | Doravirie+TAF/FTC Arm (Single Arm)
Number analyzed (Participants) | 15
CSF Unbound DORAVIRINE conc. ng/ml | 53.5 [21.3 to 115.5]

8. Primary Outcome: Unbound Doravirine Concentration CSF/Plasma Ratio
Description: Unbound Doravirine CSF/plasma ratio
Time Frame: 4 Weeks
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Doravirine+TAF/FTC Arm (Single Arm)
Number analyzed (Participants) | 15
ratio | 0.99 [0.83 to 1.17]

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Doravirine+TAF/FTC Arm (Single Arm)
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 1/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Doravirine+TAF/FTC Arm (Single Arm) (N=15)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Thoracic pain (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-06-26): https://cdn.clinicaltrials.gov/large-docs/52/NCT04079452/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-26): https://cdn.clinicaltrials.gov/large-docs/52/NCT04079452/SAP_001.pdf
  • Informed Consent Form (2019-04-10): https://cdn.clinicaltrials.gov/large-docs/52/NCT04079452/ICF_002.pdf